CLINICAL TRIAL: NCT00932282
Title: Peanut OIT & Anti-IgE: Peanut Oral Immunotherapy and Anti-IgE Treatment for Peanut Allergy {NIH R21 Combined Peanut Oral Immunotherapy and Anti-IgE: Mechanistic Studies}
Brief Title: Peanut Oral Immunotherapy and Anti-Immunoglobulin E (IgE) for Peanut Allergy
Acronym: PAIE/Xolair
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-2306
Record Dates: First submitted 2009-06-10; First posted 2009-07-03 (Estimated); Results first posted 2017-09-26 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2015-10

CONDITIONS: Peanut Hypersensitivity
Keywords: Peanut; Allergy; Hypersensitivity
MeSH Terms: conditions — Peanut Hypersensitivity; Hypersensitivity | interventions — Omalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 12 month maintenance of PnOIT (Active Comparator): Randomized subjects who will stay on the maintenance dose of oral peanut immunotherapy (PnOIT) for 12 months.
  The study has 4 phases: anti-IgE therapy before immunotherapy (Omalizumab), an initial desensitization day(s), a buildup period, and a daily home maintenance phase with a final dose of 8000mg peanut flour (~50% peanut protein). Then all subjects will be randomized to an additional 1 or 2 years (12 or 24 months) of maintenance OIT. An OFC will be performed at the end of the long-term maintenance in all groups.
  Interventions: Drug: Peanut Oral Immunotherapy; Drug: Omalizumab
- 24 month maintenance of PnOIT (Active Comparator): All subjects will be on the same intervention until Randomization. Randomized subjects who will stay on the maintenance dose of peanut oral immunotherapy (PnOIT) for 24 months.
  The study has 4 phases: anti-IgE therapy before immunotherapy (Omalizumab), an initial desensitization day(s), a buildup period, and a daily home maintenance phase with a final dose of 8000mg peanut flour (~50% peanut protein). Then all subjects will be randomized to an additional 1 or 2 years (12 or 24 months) of maintenance OIT. An OFC will be performed at the end of the long-term maintenance in all groups.
  Interventions: Drug: Peanut Oral Immunotherapy; Drug: Omalizumab

INTERVENTIONS:
Drug: Peanut Oral Immunotherapy — Peanut flour taken by mouth, given every day. Dose ranges from 0.2mg of peanut flour to 8000mg of peanut flour during the maintenance phase.
  Other Names: PnOIT
Drug: Omalizumab — Omalizumab (anti-IgE) will be given for 4 months prior to starting oral immunotherapy. The medication is given as a subcutaneous injection with dose based on total IgE levels and weight at the beginning of the study. This medication is given for a total of 10 months.
  Other Names: Xolair

SUMMARY:
The purpose of this study is to determine whether the addition of anti-IgE treatment will make peanut oral immunotherapy safer, more tolerable, and more effective in treating peanut allergy.

DETAILED DESCRIPTION:
The goal of this proposal is to produce a new treatment that would benefit subjects who have peanut allergy by lowering the risk of anaphylactic reactions (desensitization), and changing the peanut-specific immune response in subjects who have peanut allergy (tolerance). This project is designed to study if peanut oral immunotherapy (OIT) will desensitize subjects with peanut hypersensitivity by regulating their oral and systemic immune reactivity and cause long-term tolerance. This study will augment other ongoing studies by looking at whether anti-IgE therapy can reduce side effects and allow for an accelerated build up phase. Peanut allergic patients greater than 12 years old will undergo omalizumab (anti-IgE) treatment for 4 months prior to peanut OIT, and they will continue omalizumab until one month after maintenance therapy. Each subject will have an initial desensitization phase over 2 days to a goal of 950 mg of peanut powder followed by a build up phase over 4 months to goal maintenance dose of 8000 mg peanut powder. They will be randomized to continue maintenance for 12 or 24 months. They will then have an oral food challenge (OFC) immediately after stopping peanut OIT to test for desensitization. Four weeks later, off OIT, another food challenge will be done to assess tolerance. Outcome variables of interest include results of the OFCs, pre and post skin tests, CAP-FEIA values and basophil studies. These results will be compared between the starting point and the patient at the end of the study using appropriate statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age 12 years and above of either sex, any race, any ethnicity at the time of the initial visit
* The presence of IgE specific to peanuts (a positive skin prick test to peanuts (diameter of wheal > 3.0 mm) and a positive in vitro IgE [CAP-FEIA] > 5 kUA/L
* A history of significant clinical symptoms (urticaria, angioedema, rhinorrhea, nasal congestion, pruritis, sneezing, abdominal pain, emesis, diarrhea, wheezing, shortness of breath, lip/tongue swelling, throat itching, throat swelling, impending sense of doom) occurring within 60 minutes after ingesting peanuts
* Provide signed informed consent
* Women who are sexually active, must agree to use appropriate contraceptive measures for the duration of the study and for 9 months afterwards

Exclusion Criteria:

* History of severe anaphylaxis to peanut or omalizumab as defined by hypoxia, hypotension, or neurological compromise (Cyanosis or oxygen saturation < 92% at any stage, hypotension, confusion, collapse, loss of consciousness; or incontinence)
* Currently participating in a study using an investigational new drug
* Participation in any interventional study for the treatment of food allergy in the past 12 months
* Subjects with a known oat or wheat (because of potential cross contamination with oat) food allergy will be excluded
* Poor control or persistent activation of atopic dermatitis
* Moderate to severe persistent asthma
* Currently being treated with greater than medium daily doses of inhaled corticosteroids, as defined by the National Heart Lung and Blood Institute (NHLBI) guidelines
* Inability to discontinue antihistamines for skin testing and oral food challenges (OFCs)
* History of other serious underlying disease (i.e., heart disease, diabetes, etc.)
* Women who are pregnant or nursing

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-07; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wesley Burks, MD, Principal Investigator — University of North Carolina
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 12 Month Maintenance of PnOIT: Subjects randomized to receive maintenance oral peanut immunotherapy (PnOIT) for 12 months prior to the desensitization food challenge.
- 24 Month Maintenance of PnOIT: Subjects randomized to receive maintenance oral peanut immunotherapy (PnOIT) for 24 months prior to the desensitization food challenge.
Period: Pre-OIT Anti-IgE Therapy Phase
Arm/Group | 12 Month Maintenance of PnOIT | 24 Month Maintenance of PnOIT
Started | 7 | 6
Completed | 6 | 5
Not Completed | 1 | 1
Period: Modified OIT Rush Desensitization Phase
Arm/Group | 12 Month Maintenance of PnOIT | 24 Month Maintenance of PnOIT
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0
Period: Biweekly OIT Buildup Phase
Arm/Group | 12 Month Maintenance of PnOIT | 24 Month Maintenance of PnOIT
Started | 6 | 5
Completed | 5 | 4
Not Completed | 1 | 1
Period: OIT Maintenance Phase
Arm/Group | 12 Month Maintenance of PnOIT | 24 Month Maintenance of PnOIT
Started | 5 | 4
Completed | 4 | 2
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 12 Month Maintenance of PnOIT | 24 Month Maintenance of PnOIT | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 6 | 12
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 14.4 [12.6 to 19.9] | 14.1 [12.8 to 16.1] | 14.4 [12.6 to 19.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 4 | 3 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Subjects Who Pass the 20gm Peanut Flour (~50% Peanut Protein) Oral Food Challenge 2-4 Weeks After Discontinuing Peanut OIT Therapy
Description: The primary efficacy outcome of the study is to evaluate whether the addition of anti-IgE therapy using Xolair to peanut oral immunotherapy is able to induce clinical tolerance as measured by passing an oral food challenge to 20 grams of peanut flour, 2-4 weeks after discontinuing peanut OIT therapy
Time Frame: approximately 24 or 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | 12 Month Maintenance of PnOIT | 24 Month Maintenance of PnOIT
Number analyzed (Participants) | 7 | 6
Participants | 3 | 1

2. Secondary Outcome: The Percentage of Subjects Who Tolerate the Initial Desensitization Day(s) to 950mg of Peanut Flour.
Description: A secondary efficacy outcome of the study is to evaluate whether the addition of anti-IgE therapy using Xolair to a peanut oral immunotherapy protocol allows for a higher amount of peanut tolerated after the rush desensitization phase, thereby reducing the duration of buildup phase and achieving maintenance dosing more rapidly
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | 12 Month Maintenance of PnOIT | 24 Month Maintenance of PnOIT
Number analyzed (Participants) | 7 | 6
Participants | 1 | 2

3. Secondary Outcome: The Percentage of Subjects Who Pass the 20gm Peanut Flour (~50% Peanut Protein) Oral Food Challenge Following the Desensitization Phase of the Study
Description: A secondary efficacy outcome of the study is to evaluate whether the addition of anti-IgE therapy using Xolair to peanut oral immunotherapy is able to induce clinical desensitization as measured by passing an oral food challenge to 20 grams of peanut flour on the final day of peanut OIT dosing.
Time Frame: approximately 24 or 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | 12 Month Maintenance of PnOIT | 24 Month Maintenance of PnOIT
Number analyzed (Participants) | 7 | 6
Participants | 4 | 2

4. Secondary Outcome: Incidence of All Serious Adverse Events During the Study
Description: A secondary safety outcome of the study is to determine the frequency of SAEs during oral immunotherapy in order to assess whether the addition of anti-IgE therapy using Xolair to peanut oral immunotherapy can reduce the number of SAEs that occur during oral immunotherapy when compared to previously published results
Time Frame: approximately 24 or 36 months
Measure: Number; unit: SAEs per 100 OIT doses taken
Arm/Group | 12 Month Maintenance of PnOIT | 24 Month Maintenance of PnOIT
Number analyzed (Participants) | 7 | 6
SAEs per 100 OIT doses taken | 0 | 0

5. Secondary Outcome: Incidence of Side Effects During Initial Escalation and Build up Phase of Peanut Oral Immunotherapy
Description: The primary safety outcome of the study is to determine the frequency of side effects during oral immunotherapy in order to assess whether the addition of anti-IgE therapy using Xolair to peanut oral immunotherapy can reduce the number of allergic symptoms that occur during oral immunotherapy when compared to previously published results
Time Frame: approximately 24 or 36 months
Measure: Number; unit: side effects reported per 100 OIT doses
Arm/Group | 12 Month Maintenance of PnOIT | 24 Month Maintenance of PnOIT
Number analyzed (Participants) | 7 | 6
side effects reported per 100 OIT doses | 2.8 | 3.0

ADVERSE EVENTS:
Time Frame: AE data collected over approximately 24-36 months depending on patient randomization
Arm/Group | 12 Month Maintenance of PnOIT | 24 Month Maintenance of PnOIT
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 4/7 | 3/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 12 Month Maintenance of PnOIT (N=7) | 24 Month Maintenance of PnOIT (N=6)
Vomiting (Gastrointestinal disorders) | 2 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 0
Erythematous rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Oropharyngeal itching (Skin and subcutaneous tissue disorders) | 3 | 2
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nose itch (Respiratory, thoracic and mediastinal disorders) | 0 | 0
Skin itch (Skin and subcutaneous tissue disorders) | 2 | 1
Eye or lip swelling (Skin and subcutaneous tissue disorders) | 0 | 0
Eye itch (Eye disorders) | 0 | 0
Eye tearing (Eye disorders) | 0 | 0
Hives (Skin and subcutaneous tissue disorders) | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No